CLINICAL TRIAL: NCT03383016
Title: Interaction Between Environment, Diet, Physical Activities, and Sexual Habits, in the Risk of Prostate Cancer. Validation of Biomarkers to Personalize Preventive Interventions (BIOCaPPE)
Brief Title: Diet, Physical Activity and Related Candidate Biomarkers in Relation to Prostate Cancer Risk (BIOCaPPE)
Acronym: BIOCaPPE
Status: Active, not recruiting | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: PCa19; GRéPEC-17409 (Other Grant/Funding Number: Cancer Research Society & FRQ-S)
Record Dates: First submitted 2017-12-05; First posted 2017-12-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Epidemiology; Prostate Cancer
Keywords: Prostate cancer risk; Environmental risk factors; Biomarkers; Inflammation and prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, whole blood and blood DNA samples and excess tissue collected from prostate biopsy or prostate surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men at high-rik of prostate cancer: Lifestyle questionnaires such as diet questionnaire, physical activities questionnaires, quality of life , Follows up 1 year and 2 years after the enrollment, Anthropometric measures during the first visit , Blood withdrawal for laboratory biomarkers analysis After 2 years, proposal for a 2-year end-of-study prostate biopsy to assess the presence or absence of prostate cancer.
  Interventions: Other: Lifestyle questionnaires; Diagnostic Test: Prostate Biopsy

INTERVENTIONS:
Other: Lifestyle questionnaires
  Other Names: Blood withdrawal for Laboratory biomarkers analysis; Anthropometric measures
Diagnostic Test: Prostate Biopsy — Possible follow-up by an urologist at 1 year and 2 years after recruitment. After 2 years, proposal for a 2-year end-of-study prostate biopsy to assess the presence or absence of prostate cancer.
  Other Names: follow-up by an urologist

SUMMARY:
The risk of prostate cancer is associated with lifestyle habits, such as diet and physical activity. Indeed, results of numerous studies suggest links between obesity, diabetes, inflammation and androgen and estrogen metabolism in the pathogenesis of prostate cancer.

The goal of BIOCaPPE study (Biomarkers and Prostate Cancer/ Prevention and Environment) is to identify biomarkers of prostate cancer risk that are potentially modifiable by environmental exposures (e.g. diet and physical activity).

A selection of few of the most promising biological markers will be evaluated in a cohort of more than 2000 men at high-risk of prostate cancer.

Such biomarkers would provide a practical approach to identify men at high risk of prostate cancer who could benefit from interventions aiming at reducing their risk. The biomarkers would also be useful to monitor the efficacy of the interventions on patient's lifestyle.

DETAILED DESCRIPTION:
The main objective of the proposed research project is to assess the association between five candidate biological markers potentially modifiable by environmental exposures (diet and physical activity) and the two-year risk of prostate cancer in a newly recruited cohort of men at high-risk of prostate cancer showing no evidence of cancer.

Four hospitals in the province of Quebec (Canada) participate to the recruitment of 2,055 men at high-risk for prostate cancer, i.e. men who had a first negative prostate biopsy or whose Prostatic Specific Antigen (PSA) level is between 2.5 and 10 ng/mL without previous prostate biopsy.

The candidate biomarkers that will be tested are:

1. The ratio of ω-3/ ω-6 fatty acid content of red blood cell membranes,
2. Oxidized low density lipoprotein cholesterol
3. Adiponectin
4. Insulin growth factor-1
5. The ratio of dihydrotestosterone glucuronide derivatives over estradiol

A biobank, composed of biological material (whole blood, plasma, serum, lymphocyte layer and excess tissue collected from prostate biopsy or prostate surgery) and clinical data is being created. Questionnaires are used to compile information on socio-demographic aspects, family and personal medical history, quality of life, lifestyle like food and sexual habits.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: A first negative prostate biopsy within 6 months
* Group 2: serum-PSA level between 2.5-10 ng/mL and no prior prostate biopsy

Exclusion Criteria:

* Prostate cancer
* Positive result for transurethral prostatic resection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants for this prospective cohort study are men at risk for prostate cancer.
Sampling Method: Probability Sample
Enrollment: 2053 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Biomarkers and modifiable exposure environment | An average of 2 years
  Assess the association between five candidate biological markers potentially modifiable by environmental exposures, mainly diet and physical activity, with the two-year risk of prostate cancer in men at risk for prostate cancer as previously defined.

SECONDARY OUTCOMES:
Study biobank | Through study completion, every year up to 2 years
  Biobank of biological samples, clinical data and data from the lifestyle questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Vincent FRADET, MD, PhD, Principal Investigator — CHU de Québec-Université Laval
Locations (4):
- Canada (4):
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CHU de Quebec- Université Laval, Québec, Quebec
  - Centre de recherche du Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided